CLINICAL TRIAL: NCT00532948
Title: A Phase I Trial of Capecitabine Rapidly Disintegrating Tablets and Concomitant Radiation Therapy in Children With Newly Diagnosed Brainstem Gliomas and High Grade Gliomas
Brief Title: A Study of Xeloda (Capecitabine) Plus Radiation Therapy in Children With Newly Diagnosed Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO18517
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-10

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Capecitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: capecitabine [Xeloda]

INTERVENTIONS:
Drug: capecitabine [Xeloda] — 500mg/m2 po bid (starting dose)

SUMMARY:
This single arm study will assess the maximum tolerated dose, and dose-limiting toxicities, of Xeloda administered concurrently with radiation therapy, in children with newly diagnosed diffuse intrinsic brain stem gliomas and high grade gliomas. Xeloda will be administered twice daily, at a starting dose of 500mg/m2 bid, beginning within 24 hours of the start of radiation therapy. Subsequent dose escalations will be in increments of 30%, using a standard dose escalation schema. Post-radiation therapy with Xeloda will continue after a 2 week break. The anticipated time on study treatment is 3-12 months, and the target sample size will not exceed 30 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* patients >=3 and <=21 years of age;
* newly diagnosed non-disseminated brainstem glioma or non-disseminated high grade glioma;
* Karnofsky (if >16 years) or Lansky (if < 16 years) Performance Scale of >=50%;
* adequate organ function.

Exclusion Criteria:

* previous chemotherapy, radiation therapy, immunotherapy or bone marrow transplant;
* uncontrolled infection;
* known DPD deficiency.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2007-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (9):
- United States (9):
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants in the study were enrolled at Pediatric Brain Tumor Consortium (PBTC) institutions in the United States of America (USA), from 24 May 2007 through 27 October 2009.
Pre-assignment Details: The study consisted of two periods of dosing: A dose-finding treatment period of 11 weeks and a post radiation treatment phase that lasted for 9 weeks.
Groups:
- Capecitabine 500 mg/m^2: Capecitabine 500 mg/m^2 was administered twice daily for 14 days, followed by 7 day rest. Treatment was administered for three cycles with radiation therapy period and 3 cycles without radiation therapy.
- Capecitabine 650 mg/m^2: Capecitabine 650 mg/m^2 was administered twice daily for 14 days, followed by 7 day rest. Treatment was administered for three cycles with radiation therapy period and 3 cycles without radiation therapy.
- Capecitabine 850 mg/m^2: Capecitabine 850 mg/m^2 was administered twice daily for 14 days, followed by 7 day rest. Treatment was administered for three cycles with radiation therapy period and 3 cycles without radiation therapy.
Period: Overall Study
Arm/Group | Capecitabine 500 mg/m^2 | Capecitabine 650 mg/m^2 | Capecitabine 850 mg/m^2
Started | 4 | 14 | 6
Completed | 0 | 9 | 2
Not Completed | 4 | 5 | 4
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Death | 3 | 3 | 4
Not completed — Violation of selection criteria at entry | 0 | 1 | 0
Not completed — Failure to return | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population defined as all participants enrolled.
Groups:
- Capecitabine 500 mg/m^2: Capecitabine 500 mg/m^2 was administered twice daily (ideally administered daily in two divided doses approximately 12 hours apart beginning within 24 hours of the start of radiation therapy) for 14 days, followed by 7 day rest. Treatment was administered for three cycles with radiation therapy period and 3 cycles without radiation therapy.
- Capecitabine 650 mg/m^2: Capecitabine 650 mg/m^2 was administered twice daily (ideally administered daily in two divided doses approximately 12 hours apart beginning within 24 hours of the start of radiation therapy) for 14 days, followed by 7 day rest. Treatment was administered for three cycles with radiation therapy period and 3 cycles without radiation therapy.
- Capecitabine 850 mg/m^2: Capecitabine 850 mg/m^2 was administered twice daily (ideally administered daily in two divided doses approximately 12 hours apart beginning within 24 hours of the start of radiation therapy) for 14 days, followed by 7 day rest. Treatment was administered for three cycles with radiation therapy period and 3 cycles without radiation therapy.
- Total: Total of all reporting groups
Arm/Group | Capecitabine 500 mg/m^2 | Capecitabine 650 mg/m^2 | Capecitabine 850 mg/m^2 | Total
Number analyzed (Participants) | 4 | 14 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (1.73) | 8.4 (2.65) | 13 (3.41) | 9.37 (3.39)
Gender [Count of Participants; unit: Participants]
  Female | 1 | 12 | 2 | 15
  Male | 3 | 2 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Capecitabine.
Description: The MTD was the dose level at which six evaluable patients had been treated and at most one patient experienced a dose limiting toxicity (DLT) and the next highest dose level was too toxic. Dose escalation occurred if 0 out of 3 or at most 1 out of 6 patients experienced DLT while being treated at a dose level; otherwise the dose was declared unsafe and thus above the MTD.
Time Frame: Upto 11 weeks.
Population: The safety population consisted of all eligible patients who received at least one dose of capecitabine.
Measure: Number; unit: milligrams
Groups:
- Capecitabine (Overall): Capecitabine 500, 650, and 850 mg/m^2 was administered twice daily for 14 days, followed by 7 day rest. Treatment was administered for three cycles with radiation therapy period and 3 cycles without radiation therapy
Arm/Group | Capecitabine (Overall)
Number analyzed (Participants) | 22
milligrams | 650

2. Primary Outcome: Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any of the following events occurring during the 11 week dose-finding period: any event that leads to interruption of planned radiation for 5 consecutive days or 10 days total; Grade 4 neutropenia or thrombocytopenia; Grade 3 thrombocytopenia that required a platelet transfusion on 2 or more occasions; any Grade 3 or 4 non-hematologic toxicity (with the exception of grade 3 nausea or vomiting of less than 5 days duration, Grade 3 transaminases that returned to baseline value within 7 days of study drug interruption and that did not recur upon re-challenge with study drug, and/or Grade 3 fever or infection of <5 days duration); Grade 2 non-hematologic toxicities that persisted for >7 days and required treatment interruption, or any other capecitabine-related adverse events that required need for dose reduction or permanent cessation of therapy, interruption of study drug for >7 days or recurred on re-challenge with capecitabine rapidly disintegrating tablets (RDTs).
Time Frame: Upto 11 weeks
Population: The safety population consisted of all eligible patients who received at least one dose of capecitabine.
Measure: Number; unit: Participants
Arm/Group | Capecitabine 500 mg/m^2 | Capecitabine 650 mg/m^2 | Capecitabine 850 mg/m^2
Number analyzed (Participants) | 4 | 12 | 6
Participants | 0 | 3 | 3

3. Primary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE is an unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Toxicity was monitored and graded according to the Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Adverse events that were not included in the CTCAEv3.0 were reported and graded under the other AE within the appropriate category.
Time Frame: Up to 06 years
Population: The safety population consisted of all eligible patients who received at least one dose of capecitabine.
Measure: Number; unit: Participants
Arm/Group | Capecitabine 500 mg/m^2 | Capecitabine 650 mg/m^2 | Capecitabine 850 mg/m^2
Number analyzed (Participants) | 4 | 12 | 6
Participants | 3 | 12 | 6

4. Primary Outcome: Number of Participants With Baseline Shift From Normal to Low or High in Hematology Parameters
Description: For hematology, the parameters assessed were: Hemoglobin, hematocrit, platelet count, RBC, WBC, lymphocytes, monocytes,granulocytes (blasts), neutrophils(segs, bands),eosinophils and basophils.
Time Frame: Up to 06 years
Population: The safety population consisted of all eligible patients who received at least one dose of capecitabine. Participants available at a particular time point were included in analysis.
Measure: Number; unit: Participants
Arm/Group | Capecitabine 500 mg/m^2 | Capecitabine 650 mg/m^2 | Capecitabine 850 mg/m^2
Number analyzed (Participants) | 4 | 12 | 6
Participants
  Haematocrit, normal to low, n=3,1,5 | 2 | 1 | 4
  Haematocrit, normal to high, n=3,1,5 | 0 | 0 | 0
  Hemoglobin, normal to low, n=4,2,6 | 0 | 0 | 2
  Hemoglobin, normal to high, n=4,2,6 | 0 | 0 | 0
  White blood cell, normal to low, n=3,1,5 | 0 | 0 | 0
  White blood cell, normal to high, n=3,1,5 | 1 | 1 | 1
  Platelets, normal to low, n=4,2,6 | 0 | 1 | 0
  Platelets, normal to high, n=4,2,6 | 0 | 0 | 1
  Red blood cells, normal to low, n=3,1,3 | 2 | 0 | 1
  Red blood cells, normal to high, n=3,1,3 | 0 | 1 | 0
  Neutrophils (segmented), normal to low , n=3,0,5 | 0 | 0 | 0
  Neutrophils (segmented), normal to high, n=3,0,5 | 0 | 0 | 0
  Basophils (relative), normal to low, n=0,1,2 | 0 | 0 | 0
  Basophils (relative), normal to high, n=0,1,2 | 0 | 1 | 2
  Lymphocytes (relative), normal to low, n=3,1,5 | 0 | 0 | 0
  Lymphocytes (relative), normal to high, n=3,1,5 | 0 | 0 | 0
  Monocytes (relative), normal to low, n=3,1,4 | 0 | 0 | 0
  Monocytes (relative), normal to high, n=3,1,4 | 1 | 0 | 3
  Eosinophils (relative), normal to low, n=1,1,3 | 0 | 1 | 0
  Eosinophils (relative), normal to high, n=1,1,3 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Baseline Shift From Normal to Low or High in Blood Chemistry Parameters
Description: For blood chemistry, the parameters assessed were: Sodium, potassium, calcium, magnesium, chloride, bicarbonate, total protein, albumin, alkaline phosphatase, alanine transaminase (ALT), aspartate aminotransferase (AST), blood urea nitrogen (BUN), Lactate dehydrogenase (LDH), total bilirubin, direct bilirubin, indirect bilirubin, creatinine (serum creatinine or creatinine clearance), glucose.
Time Frame: Up to 06 years
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Capecitabine 500 mg/m^2 | Capecitabine 650 mg/m^2 | Capecitabine 850 mg/m^2
Number analyzed (Participants) | 4 | 12 | 6
Participants
  Lactic dehydrogenase, normal to low, n=0,0,0 | 0 | 0 | 0
  Lactic dehydrogenase, normal to high, n=0,0,0 | 0 | 0 | 0
  Indirect bilirubin, normal to low, n=1,1,1 | 0 | 0 | 0
  Indirect bilirubin, normal to high, n=1,1,1 | 0 | 1 | 0
  BUN, normal to low, n=3,1,5 | 0 | 0 | 2
  BUN, normal to high, n=3,1,5 | 0 | 1 | 1
  Alkaline phosphatase, normal to low, n=1,1,4 | 0 | 0 | 1
  Alkaline phosphatase, normal to high, n=1,1,4 | 0 | 0 | 0
  Direct blirubin, normal to low, n=2,1,1 | 0 | 0 | 0
  Direct bilirubin, normal to high, n=2,1,1 | 0 | 0 | 0
  Total bilirubin, normal to low, n=4,2,6 | 0 | 0 | 0
  Total bilirubin, normal to high, n=4,2,6 | 0 | 0 | 0
  Fasting glucose, normal to low, n=1,0,4 | 0 | 0 | 0
  Fasting glucose, normal to high, n=1,0,4 | 0 | 0 | 0
  Protein, normal to low, n=1,0,2 | 1 | 0 | 1
  Protein, normal to high, n=1,0,2 | 0 | 0 | 0
  Serum albumin, normal to low, n=3,1,5 | 2 | 0 | 1
  Serum albumin, normal to high, n=3,1,5 | 0 | 0 | 0
  Serum creatinine, normal to low, n=4,2,6 | 0 | 0 | 0
  Serum creatinine, normal to high, n=4,2,6 | 0 | 0 | 2
  ASAT (SGOT), normal to low, n=1,0,4 | 0 | 0 | 0
  ASAT (SGOT), normal to high, n=1,0,4 | 0 | 0 | 2
  ALAT (SGPT), normal to low, n=4,2,6 | 0 | 0 | 0
  ALAT (SGPT), normal to high, n=4,2,6 | 2 | 2 | 4
  Calcium, normal to low, n=3, 1,5 | 1 | 1 | 0
  Calcium, normal to high, n=3,1,5 | 0 | 0 | 1
  Phosphate, normal to low, n=3,1,5 | 1 | 0 | 1
  Phosphate, normal to high, n=3,1,5 | 0 | 0 | 1
  Potassium, normal to low, n=3, 1,5 | 2 | 0 | 0
  Potassium, normal to high, n=3,1,5 | 0 | 1 | 0
  Sodium, normal to low, n=3,1,5 | 1 | 1 | 3
  Sodium, normal to high, n=3,1,5 | 0 | 0 | 0
  Magnesium, normal to low, n=3,1,5 | 0 | 0 | 0
  Magnesium, normal to high, n=3,1,5 | 1 | 1 | 0
  Chloride, normal to low, n=3,1,5 | 0 | 0 | 1
  Chloride, normal to high, n=3,1,5 | 0 | 1 | 1
  Bicarbonate, normal to low, n=3,0,5 | 0 | 0 | 0
  Bicarbonate, normal to high, n=3,0,5 | 0 | 0 | 3

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Capecitabine and Its Metabolites (5'-Deoxy-5-Fluorocytidine [5'-DFCR], 5'-Deoxy-5-Fluorouridine [5'-DFUR], 5-Fluorouracil [5-FU] and Alpha-fluoro-beta-alanine [FBAL])
Description: The maximum observed plasma concentration of capecitabine and its metabolites. Participants who consented to participating in the PK studies were randomized to either sampling series A or Series B. The collection time points included 2 different series, Series A (Baseline [pre-dose], 10 mins, 30 mins, 1, 2.5, 6, 8 and 10 hours after dosing) and Series B (Baseline [pre-dose], 15 minutes, 45 minutes, 1.5, 4, 8 and 10 hours after dosing).
Time Frame: Day 1 and Day 14
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Capecitabine 500 mg/m^2 | Capecitabine 650 mg/m^2 | Capecitabine 850 mg/m^2
Number analyzed (Participants) | 4 | 6 | 5
ng/mL
  Capecitabine, Day 1, n= 2, 4, 3 | 1440 (750) | 3080 (1340) | 1890 (1420)
  Capecitabine, Day 14, n=2,2,2 | 2100 (1770) | 5440 (3270) | 3710 (156)
  5'-DFCR, Day 1, n=2,4,3 | 2050 (813) | 2190 (626) | 2180 (1690)
  5'-DFCR, Day 14, n=2,2,2 | 2980 (2020) | 3500 (1470) | 3200 (233)
  5'-DFUR, Day 1, n=2,4,3 | 1910 (834) | 2640 (1700) | 3770 (3300)
  5'-DFUR, Day 14, n=2,2,2 | 3300 (2800) | 3120 (445) | 5020 (1220)
  FBAL, Day 1, n=2,4,3 | 1350 (134) | 1740 (365) | 2050 (1640)
  FBAL, Day 14, n=2,2,2 | 1770 (410) | 2430 (84.9) | 2140 (304)

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Capecitabine and Its Metabolites (5'-DFCR, 5'-DFUR, 5-FU and FBAL)
Description: Tmax is the corresponding time at which Cmax occurs of capecitabine and its metabolites.Participants who consented to participating in the PK studies were randomized to either sampling series A or Series B. The collection time points included 2 different series, Series A (Baseline [pre-dose], 10 mins, 30 mins, 1, 2.5, 6, 8 and 10 hours after dosing) and Series B (Baseline [pre-dose], 15 minutes, 45 minutes, 1.5, 4, 8 and 10 hours after dosing).
Time Frame: Day 1 and Day 14
Population: as for outcome 4
Measure: Median (Full Range); unit: Hour
Arm/Group | Capecitabine 500 mg/m^2 | Capecitabine 650 mg/m^2 | Capecitabine 850 mg/m^2
Number analyzed (Participants) | 4 | 6 | 5
Hour
  Capecitabine, Day 1, n= 2, 4, 3 | 0.58 [0.17 to 1] | 0.63 [0.25 to 1] | 0.85 [0.83 to 10]
  Capecitabine, Day 14, n=2,2,2 | 1.33 [0.17 to 2.48] | 0.82 [0.8 to 0.83] | 0.61 [0.5 to 0.72]
  5'-DFCR, Day 1, n=2,4,3 | 1.0 [1.0 to 1.0] | 0.75 [0.50 to 2.50] | 1.55 [0.85 to 10]
  5'-DFCR, Day 14, n=2,2,2 | 1.49 [0.5 to 2.48] | 1.18 [0.5 to 1.53] | 0.61 [0.5 to 1.53]
  5'-DFUR, Day 1, n=2,4,3 | 1 [1 to 1] | 0.9 [0.7 to 2.5] | 1.5 [0.75 to 10]
  5'-DFUR, Day 14, n=2,2,2 | 1.5 [0.5 to 2.5] | 0.82 [0.8 to 0.83] | 0.61 [0.5 to 0.72]
  5-FU, Day 1, n=2,4,3 | 1 [1 to 1] | 0.75 [0.5 to 2.5] | 1.5 [0.75 to 10]
  5-FU, Day 14, n=2,2,2 | 1.5 [0.5 to 2.5] | 0.83 [0.8 to 0.83] | 1 [0.5 to 1.5]
  FBAL, Day 1, n=2,4,3 | 2.53 [2.5 to 2.53] | 1.5 [1.5 to 2.5] | 1.55 [1.42 to 10]
  FBAL, Day 14, n=2,2,2 | 1.74 [1 to 2.5] | 2.2 [1.5 to 2.8] | 2.03 [1.57 to 2.5]

8. Secondary Outcome: The Area Under the Plasma Concentration-time Curve From Time of Dosing to the Last Measurable Concentration (AUClast) of Capecitabine and Its Metabolites (5'-DFCR, 5'-DFUR, 5-FU and FBAL)
Description: AUC last concentration of capecitabine and its metabolites. Participants who consented to participating in the PK studies were randomized to either sampling series A or Series B. The collection time points included 2 different series, Series A (Baseline [pre-dose], 10 mins, 30 mins, 1, 2.5, 6, 8 and 10 hours after dosing) and Series B (Baseline [pre-dose], 15 minutes, 45 minutes, 1.5, 4, 8 and 10 hours after dosing).
Time Frame: Day 1 and Day 14
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Capecitabine 500 mg/m^2 | Capecitabine 650 mg/m^2 | Capecitabine 850 mg/m^2
Number analyzed (Participants) | 4 | 6 | 5
h*ng/mL
  Capecitabine, Day 1, n= 2, 4, 3 | 3370 (607) | 5160 (3700) | 3470 (1170)
  Capecitabine, Day 14, n=2,2,2 | 2890 (655) | 9660 (3340) | 5670 (971)
  5'-DFCR, Day 1, n=2,4,3 | 5250 (755) | 5140 (3440) | 4180 (2380)
  5'-DFCR, Day 14, n=2,2,2 | 4300 (27.2) | 9250 (1400) | 6520 (452)
  5'-DFUR, Day 1, n=2,4,3 | 4790 (784) | 4300 (1600) | 6650 (3740)
  5'-DFUR, Day 14, n=2,2,2 | 4240 (929) | 8010 (1890) | 10500 (445)
  5-FU Day 1, n=2,4,3 | 81.6 (29.7) | 114 (40.9) | 271 (205)
  5-FU Day 14, n=2,2,2 | 181 (84.7) | 253 (16.3) | 499 (78.8)
  FBAL, Day 1, n=2,4,3 | 5990 (951) | 8110 (1640) | 7010 (4490)
  FBAL, Day 14, n=2,2,2 | 5720 (690) | 10700 (574) | 10400 (1760)

9. Secondary Outcome: Anti Tumor Activity
Description: Tumor response refers to the best response prior to failure (disease progression, death or second malignancy).
Time Frame: Up to 6 years
Population: Efficacy data of the present study (NO18517 - NCT00532948) were pre-specified to be combined with efficacy data of the Phase 2 portion of this Study, NO21125 (NCT01118377) for analysis. Results are currently posted in the record of Study NO21125.
Arm/Group | Capecitabine 500 mg/m^2 | Capecitabine 650 mg/m^2 | Capecitabine 850 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 years
Arm/Group | Capecitabine 500 mg/m^2 | Capecitabine 650 mg/m^2 | Capecitabine 850 mg/m^2
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/12 | 3/6
Other Adverse Events (participants affected / at risk) | 3/4 | 12/12 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine 500 mg/m^2 (N=4) | Capecitabine 650 mg/m^2 (N=12) | Capecitabine 850 mg/m^2 (N=6)
Convulsion (Nervous system disorders) | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Abdominal Infection (Infections and infestations) | 0 | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine 500 mg/m^2 (N=4) | Capecitabine 650 mg/m^2 (N=12) | Capecitabine 850 mg/m^2 (N=6)
Alanine aminotransferase increased (Investigations) | 1 | 9 | 3
Haemoglobin (Investigations) | 1 | 4 | 2
Neutrophil count (Investigations) | 2 | 4 | 1
Platelet count decreased (Investigations) | 2 | 5 | 0
Weight increased (Investigations) | 1 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1
Blood bicarbonate decreased (Investigations) | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 3 | 10 | 3
Leukopenia (Blood and lymphatic system disorders) | 3 | 10 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 9 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 4
Nausea (Gastrointestinal disorders) | 1 | 2 | 4
Constipation (Gastrointestinal disorders) | 1 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 8 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 4 | 2
Convulsion (Nervous system disorders) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 2 | 0
VIth nerve disorder (Nervous system disorders) | 1 | 2 | 0
Ataxia (Nervous system disorders) | 1 | 1 | 0
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Otitis media (Infections and infestations) | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 2 | 1
Hypertension (Cardiac disorders) | 1 | 2 | 0
Diplopia (Eye disorders) | 2 | 0 | 0
Extraocular muscle disorder (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Euphoric mood (Psychiatric disorders) | 0 | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 1
Oculomotor nerve operation (Surgical and medical procedures) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.